CLINICAL TRIAL: NCT04491409
Title: ARCA-1 Study: Perioperative Care in the Cancer Patient -1
Brief Title: Perioperative Care in the Cancer Patient -1, ARCA-1 Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0130; NCI-2020-04546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0130 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-14; First posted 2020-07-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (standard of care, medical chart review): Patients undergo standard of care treatment and their medical records are reviewed at 30 days and at 1 year after surgery.
  Interventions: Other: Best Practice; Other: Medical Chart Review

INTERVENTIONS:
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
Other: Medical Chart Review — Medical charts reviewed
  Other Names: Chart Review

SUMMARY:
This study investigates the association of blood transfusions given around the time of surgery (perioperative) with complications after surgery (postoperative), cancer progression, and mortality after major oncologic non-cardiac surgery. The administration of blood products is an important clinical therapy to treat life-threatening blood (hematological) disorders (i.e. anemia, coagulation disorders or thrombocytopenia) in patients with cancer undergoing major non-cardiac surgery. On the other hand, the unnecessary exposure of those patients to blood products can be associated with the occurrence of unwanted severe complications and potentially increase the risk of death. An accurate understanding of the short and long-term outcomes, the patterns of blood transfusions, and the triggers of blood product administration may help researchers design and test the safety of perioperative blood transfusions in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if perioperative blood transfusions are associated with 1-year mortality.

SECONDARY OBJECTIVES:

I. To evaluate the association of blood transfusion with postoperative complications, 30 days mortality and cancer progression after major oncologic non-cardiac surgery.

II. To gain knowledge on prevalence and patterns of blood product administration worldwide, the incidence and management of perioperative anemia and the incidence and treatment of perioperative coagulopathies.

OUTLINE:

Patients undergo standard of care treatment and their medical records are reviewed at 30 days and at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major cancer surgery with curative intent
* Planned length of stay 24 hours after surgery or longer
* American Society of Anesthesiologists physical status (ASA) 1-4
* Scheduled, non-emergency surgery

Exclusion Criteria:

* Emergency surgery
* Palliative surgeries for metastatic disease (non-curative intent)
* Patients undergoing surgery with minimum risk (< 1%) of blood transfusion according to each center practice (i.e. simple mastectomy, thyroidectomies or wide-local excisions)
* Patients undergoing surgery under local anesthesia
* Patients undergoing ambulatory surgery or planned hospital admission of less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing major cancer surgery with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
All causes of mortality | 1 year after major oncologic non-cardiac surgery

SECONDARY OUTCOMES:
Cancer-specific mortality | 1 year after major oncologic non-cardiac surgery
Progression free survival (PFS) | From the date of surgery to the date of progression or death whichever happened first, assessed at 1 year after major oncologic non-cardiac surgery
  Kaplan-Meier method will be used to estimate the PFS, and the log-rank test will be used to evaluate the difference in PFS between the RBCT group and non-RBCT group. PFS rate at 1 year will be reported. Multivariable Cox proportional hazards models may be used to evaluate the effect of RBCT on PFS with the adjustment of other important covariates.
30 days mortality | 30 days after major oncologic non-cardiac surgery
Rate of perioperative blood products transfusion | During surgery and up to 2 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Cata, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cata JP, Guerra-Londono JJ, Ramirez MF, Chen LL, Warner MA, Guzman LFC, Lobo F, Uribe-Marquez S, Huang J, Ruscic KJ, Chew STH, Lanigan M; ARCA-1 Investigators. The Association Between Perioperative Red Blood Cell Transfusions and 1-Year Mortality After Major Cancer Surgery: An International Multicenter Observational Study. Anesth Analg. 2025 Apr 1;140(4):782-794. doi: 10.1213/ANE.0000000000007236. Epub 2024 Nov 6. PMID 39504267
- [Derived] Cata J, Ramirez M, Forget P, Chen LL, Diaz-Cambronero O, Chen W, Warner MA, Knopfelmacher Couchonal A, Pelosi P, Cuellar L, Corrales G, Romero C, Lobo F, Saager L, Castro Tapia J, Kiberenge R, Feng L, Serpa Neto A. International multicentre observational study to evaluate the association between perioperative red blood cell transfusions and 1-year mortality after major cancer surgery (ARCA-1): study design, statistical analysis plan and study protocol. BMJ Open. 2021 Mar 18;11(3):e043453. doi: 10.1136/bmjopen-2020-043453. PMID 33737431
- See also: Related Info — http://www.mdanderson.org